CLINICAL TRIAL: NCT04158882
Title: Analysis of Existing Medical Record Data to Evaluate Coverage, Uptake, Benefits, and Costs of Differentiated Models of Service Delivery for HIV Treatment in Africa (Zambia)
Brief Title: Gathering Records to Evaluate Antiretroviral Treatment-Zambia (GREAT )
Acronym: GREAT
Status: Recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Witwatersrand, South Africa (Other); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: H-38823
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HIV
Keywords: HIV; Zambia; Differentiated service delivery; Antiretroviral therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients enrolled in differentiated service delivery models
  Interventions: Other: Routine medical record data collection
- Patients not enrolled in DSD models
  Interventions: Other: Routine medical record data collection

INTERVENTIONS:
Other: Routine medical record data collection — The study will collect routine medical record data from the electronic medical record system, other electronic databases, and paper charts.

SUMMARY:
To achieve global goals for the treatment of HIV, most high-prevalence countries are experimenting with and scaling up differentiated service delivery models (DSD). A handful of efforts have been formally described and evaluated in the literature; many others are being implemented formally or informally under routine care, without a research or evaluation goal. For most countries, however, there is little evidence on the big picture-the proportion of clinics offering alternative models, eligibility criteria and the proportion of patients considered eligible, the number of patients actually participating, health outcomes such as viral suppression, empirical resource utilization compared to traditional care, variations among the models, duration of patient participation, fidelity to model guidelines, effects on clinic efficiency, and sustainability without external donor support.

AMBIT a set of data synthesis, data collection, and data analysis activities aimed at generating information for near- and long-term decision making and creating an approach and platform for ongoing evaluation of differentiated models of HIV treatment delivery in the future. The project will collect and analyze a wide range of existing data sets pertinent to DSD. This protocol is for an analysis of existing medical record data collected by the Ministry of Health, implementing partners, and other completed, ongoing, or new evaluations, trials, and observational studies. Outcomes to be reported include coverage/uptake of DSD, patients' outcomes, and distribution of each model. There will be no study interaction with individual patients, providers, caregivers, or others for this analysis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 15 years old
* Patients accessing care for HIV within the data collection period
* In any HIV transmission risk group

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adults who are accessing care for HIV anywhere in the country.
Sampling Method: Non-Probability Sample
Enrollment: 1200000 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-months enrolled in any DSD model | 12 months
  % of all patient-months of ART provided for the cohort that are provided within DSD models
Patient-months enrolled in any DSD model | 24 months
  % of all patient-months of ART provided for the cohort that are provided within DSD models
Patient-months enrolled in any DSD model | 6 months
  % of all patient-months of ART provided for the cohort that are provided within DSD models

CONTACTS AND LOCATIONS:
Overall Officials: Sydney B Rosen, Study Director — Boston University School of Pubic Health
Locations (1):
- All clinics, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jamieson L, Rosen S, Phiri B, Grimsrud A, Mwansa M, Shakwelele H, Haimbe P, Mukumbwa-Mwenechanya M, Lumano-Mulenga P, Chiboma I, Nichols BE. How soon should patients be eligible for differentiated service delivery models for antiretroviral treatment? Evidence from a retrospective cohort study in Zambia. BMJ Open. 2022 Dec 22;12(12):e064070. doi: 10.1136/bmjopen-2022-064070. PMID 36549722